CLINICAL TRIAL: NCT01001585
Title: Anesthetic Effects in Mitochondrial Disease
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: However, no intervention reduced the risk of major morbidity or 1 yr mortality
Sponsor: d sessler (Other)
Responsible Party: Sponsor-Investigator, d sessler, Medical Doctor, The Cleveland Clinic
Organization: The Cleveland Clinic (Other)
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Supportive Care
Other Study IDs: 06-644
Record Dates: First submitted 2009-10-21; First posted 2009-10-26 (Estimated); Last update posted 2015-03-09 (Estimated); Status verified 2015-03

CONDITIONS: Mitochondrial Disease
Keywords: mitochondrial disease; sevoflurane; mitochondrial disease and sevoflurane sensitivity
MeSH Terms: conditions — Mitochondrial Diseases | interventions — Sevoflurane

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- slow induction with sevoflurane (Experimental): Only children with a BIS greater than 95 prior to inhalation of sevoflurane will be included in the study. Inductions will be done using a tight fitting mask with continuous monitoring of end tidal gas concentrations. During induction, concentration of inspired sevoflurane will begin at .5%, and slowly increased by 0.5% every two minutes, until a Bispectral Index (BIS) of 60 or less is reached. Inspired sevoflurane will be increased only after end tidal concentration of sevoflurane is constant for at least one minute. Each induction (except for the patients requiring very low doses of sevoflurane) will take approximately 10 minutes.
  Interventions: Drug: sevoflurane

INTERVENTIONS:
Drug: sevoflurane — During induction, concentration of inspired sevoflurane will begin at .5%, and slowly increased by 0.5% every two minutes, until a Bispectral Index (BIS) of 60 or less is reached, which will take approximately 10 minutes.

SUMMARY:
Summary. At the present, the investigators do not have the perfect anesthetic for mitochondrial patients. When possible, consideration should be given to the use of local anesthetics in small amounts. When a general anesthetic is necessary, they each carry significant risks and have been associated with poor outcomes. At present it is not possible to eliminate one group as less safe than others. What is clear is that these patients must be monitored more closely than other patients. The advent of the bispectral index (BIS) monitor may allow us to monitor their depth of anesthesia more closely and thus expose these patients only to the minimum amount of drug necessary to carry out the surgical procedure.

Purpose. The investigators hypothesize that specific mitochondrial diseases, in particular those that decrease complex I function, make certain children hypersensitive to volatile anesthetics. These same patients may be at increased risk for adverse outcomes following general anesthesia. The specific aims of this application are:

1. Determine which molecular defects in mitochondrial function lead to alter sensitivity to the VA sevoflurane.
2. Establish the relative safety of sevoflurane in treatment of patients with mitochondrial disease.

The investigators plan to monitor patients with mitochondrial disease using expanded measures of cardiovascular stability and measurements of brain electrical activity while slowly inducing general anesthesia. The investigators will use those measurements to limit the amount of anesthetic these patients receive in an attempt to minimize their risk. In addition, the investigators will correlate their sensitivity to the type of mitochondrial defect so that the investigators may be able to predict which patients are likely to have an increased sensitivity.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting to the operating room for muscle biopsy as part of their diagnostic workup for possible mitochondrial disease.

Exclusion Criteria:

* Patients more than 16 years of age.
* Patients with concurrent acute infectious disease.
* Patients not tolerating a slow induction for emotional reasons.
* Initial BIS measurement of less than 95.
* Documented pulmonary disease.

Ages: 12 Months to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 55 (Actual)
Dates: Start 2006-09; Primary Completion 2011-09 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Measure cardiovascular stability and electrical brain activity during slow induction with sevoflurane. | during induction
  The investigators plan to monitor patients with mitochondrial disease using expanded measures of cardiovascular stability and measurements of brain electrical activity while slowly inducing general anesthesia. The investigators will use those measurements to limit the amount of anesthetic these patients receive in an attempt to minimize their risk.

SECONDARY OUTCOMES:
Use cardiovascular and electrical brain measurements to limit amount of sevoflurane and predict individual sensitivity. | during induction
  In addition, the investigators will correlate their sensitivity to the type of mitochondrial defect so that it may be possible to predict which patients are likely to have an increased sensitivity.

CONTACTS AND LOCATIONS:
Overall Officials: Danield I Sessler, MD, Study Chair — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States